CLINICAL TRIAL: NCT02911675
Title: Assessing the Accuracy and the Impact of Standard-practice Ventricular Drainage on Intracranial Pressure Measurements Following Traumatic Brain Injury
Acronym: Dual ICP
Status: Withdrawn | Type: Observational
Why Stopped: Due to the lack of approval from the Air Force IRB patient enrollment was never initiated. Thus, no clinical results could be examined or can be reported
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: United States Air Force (U.S. Federal Agency)
Responsible Party: Principal Investigator, Deborah Stein, Medical Director, Neurotrauma Critical Care; Chief, Section of Trauma Critical Care, R Adams Cowley Shock Trauma Center, University of Maryland, Baltimore
Other Study IDs: HP-00064113
Record Dates: First submitted 2016-08-24; First posted 2016-09-22 (Estimated); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Traumatic Brain Injury
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Standard of Care Group: Study Group 1: Standard EVD/IVC management with therapeutic CSF drainage as appropriate and hourly EVD/IVC ICP measurements per standard of care with simultaneous IPM/Camino ICP measurements collected.
  Interventions: Device: EVD/IVC and the IPM/Camino
- Experimental Group: Study Group 2: Therapeutic CSF drainage as appropriate, with EVD/IVC closure and ICP assessment approximately every 12 hours with simultaneous IPM/Camino ICP measurements collected.
  Interventions: Device: EVD/IVC and the IPM/Camino

INTERVENTIONS:
Device: EVD/IVC and the IPM/Camino — This is an interventional device study utilizing the EVD/IVC and the IPM/Camino to provide and evaluate data for optimized treatment for the control of elevated ICP and CCP in patients with severe TBI.

SUMMARY:
Traumatic brain injury (TBI) is a leading cause of death following injury in civilian populations and is a major cause of death and disability in combat casualties. While primary brain injury cannot be reversed, the management of severe TBI focuses on the mitigation of secondary injury mechanisms which occur as part of the downstream effects of the primary damage to the brain. Many secondary injury mechanisms are manifested clinically as elevated intracranial pressure (ICP) and cerebral perfusion pressure (CCP). This level and duration of elevated ICP is strongly associated with poor long term patient outcome.

Currently, there are two invasive techniques that are used at our facility for monitoring ICP and CPP. The first method requires the placement of an intra-parenchymal fiberoptic pressure monitor (IPM), also known as a camino, into the brain tissue that measures and displays ICP continuously. The second method requires placement of an extracranial ventricular drain (EVD) which both measures ICP when it is closed or clamped and also allows for therapeutic drainage of cerebral spinal fluid (CFS) to reduce pressure within the skull when it is open.

While clinical practices vary greatly across institutions, current clinical practice at our institution when using the EVD for ICP management is to allow continuous therapeutic CSF drainage and to manually close the drain for ICP assessment on an hourly basis. However, in a retrospective of study of TBI patients at our institution with simultaneous IPM and EVD placement, a spike in ICP was noted to correspond with the clamping of the EVD which often remained elevated for 15-30 minutes before returning to baseline. Due to the strong association between poor patient outcome and elevated ICP, this finding is alarming. These findings have important implications for procedures to not only treat elevated ICP, but also prevent potentially harmful intermittent elevations in ICP. Therefore, this study seeks to prospectively investigate the association between EVD clamping and elevated ICP.

Specifically, this study has 2 main objectives:

1. Evaluate the need for an optimized device that can simultaneously measure intracranial pressure and drain CSF without requiring potentially harmful clamping.
2. Provide data in support of retaining or modifying current clinical practices regarding intermittent versus continuous monitoring during periods of therapeutic drainage of CSF.

DETAILED DESCRIPTION:
Investigators plan a single-center, 36 month prospective observational study of 50 patients presenting with moderate to severe traumatic brain injury (TBI) at R Adams Cowley Shock Trauma Center who require intracranial pressure monitoring. This is an interventional device study utilizing the EVD/IVC and the IPM/Camino to provide and evaluate data for optimized treatment for the control of elevated ICP and CCP in patients with severe TBI. Enrolled patients will be randomized to one of two study groups listed below following the consent process. Once a potential participant has consented to the study, we will use the excel random number generator function (randbetween(0,1)) to generate random numbers between 0 and 1 for each participant. If 0 is generated participants will be placed in Group 1 (Hourly EVD closures) and if 1 is generated, participants will be placed in Group 2 (EVD closure every 12 hours). There is no placebo or control group.

Standard of Care (25 patients): Standard EVD management with therapeutic drainage as appropriate and hourly EVD ICP measurements with simultaneous IPM/Camino ICP measurements collected.

Experimental (25 patients): Therapeutic CSF drainage as appropriate, with EVD closure and ICP assessment every 12 hours with simultaneous IPM/Camino ICP measurements collected.

Data will be collected on age, mechanism of injury, time interval between injury and MRI, past medical history, admission hemodynamics, admission component GCS, post-resuscitation component GCS, injury severity score, abbreviated injury score for head injury, blunt carotid or vertebral artery injury, and therapeutic interventions. Continuous vital signs streams will be collected.

In addition, if available, video surveillance from the patient's stay in the Neurotrauma Critical Care Unit will be collected and be stored with the patients study data.

ELIGIBILITY:
Inclusion Criteria:

* Direct trauma admission to STC by ambulance or helicopter
* 18 years and older
* Neurosurgical evaluation indicates placement of a EVD
* Diagnosis of severe traumatic brain injury (head AIS > 2) and post-resuscitation motor CGS<6

Exclusion Criteria:

* < 18 years of age
* Non-survivable brain injury
* Non-survivable anatomic injury
* Pregnancy
* Non-English speaker
* Prisoner
* Active duty military

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an interventional device study utilizing the EVD/IVC and the IPM/Camino to provide and evaluate data for optimized treatment for the control of elevated ICP and CCP in patients with severe TBI. Enrolled patients will be randomized to one of two study groups listed below following the consent process. Once a potential participant has consented to the study, we will use the excel random number generator function (randbetween(0,1)) to generate random numbers between 0 and 1 for each participant. If 0 is generated participants will be placed in Group 1 (Hourly EVD closures) and if 1 is generated, participants will be placed in Group 2 (EVD closure every 12 hours). There is no placebo or control group.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-01-24 (Actual); Study Completion 2019-01-24 (Actual)

PRIMARY OUTCOMES:
Evaluate the need for an optimized device that can simultaneously measure intracranial pressure and drain CSF without requiring potentially harmful clamping. | 6 months
  Investigators want to find a better device that can measure pressure in the head after a traumatic brain without causing an increase in pressure inside of the head.

SECONDARY OUTCOMES:
Compare clinical practices regarding intermittent versus continuous monitoring during periods of therapeutic drainage of CSF. | 6 months
  Compare the current method of clamping the drain with the experimental method to determine if clamping the drain less will provide an accurate measure of pressure inside of the head.

OTHER OUTCOMES:
Evaluate the impact of the frequency of EVD drain closure on short and long (6 month) term functional outcomes. | 6 months
  Assess the impact of the frequency of EVD drain closure on short and long (6 month) term functional outcomes.

IPD SHARING:
Plan to Share IPD: No